Official Title: A Phase II Study of Optune (NovoTTF) in Combination With Bevacizumab (BEV) and Temozolomide (TMZ) in Patients With Newly Diagnosed Unresectable Glioblastoma (GBM)

NCT02343549

IRB-Approved Date: 3/7/2018

# CAROLINAS HEALTHCARE SYSTEM CONSENT TO PARTICIPATE IN A RESEARCH STUDY

Sponsor / Study Title: Levine Cancer Institute, A Phase II Study of Optune TM in

Combination with Bevacizumab (BEV) and Temozolomide (TMZ) in Patients with Newly Diagnosed, Unresectable

Glioblastoma (GBM)

Protocol Number: LCI-NEU-NOV-001

Principal Investigator: Ashley Sumrall, MD

Telephone: (24 Hours)

(24 Hours Toll Free)

Address: Levine Cancer Institute

### **INTRODUCTION**

Dr. Ashley Sumrall and her associates are asking you to participate in this research study of Optune<sup>TM</sup> and bevacizumab at Levine Cancer Institute (LCI) and Carolinas HealthCare System (CHS). You are being asked to take part because you are 22 years of age or older and have a newly diagnosed, unresectable glioblastoma (GBM). The purpose of this study is find out if using Optune<sup>TM</sup> will improve survival.

Temozolomide (TMZ) is a chemotherapy drug that is currently approved by the FDA for use in newly diagnosed GBM patients (like you). Bevacizumab (BEV) is a chemotherapy drug that is currently Food and Drug Administration (FDA) approved for use in GBM that has progressed. Optune TM in combination with BEV and TMZ is considered investigational and is not FDA approved.

You will be one of approximately 46 people involved in this research project at CHS. Your participation will last until your disease gets worse, you no longer wish to participate, or your study doctor removes you from the study.

This is a clinical trial, a type of research study. Your study doctor will explain the clinical trial to you. Clinical trials include only people who choose to take part. Please take your time to make your decision about taking part. You have also been told that you have the option not to participate. You

Ashley Sumrall, MD

Chesapeake IRB Approved Version 7 Mar 2018



Affix Participant Barcode Label Here

may discuss your decision with your friends and family. You can also discuss it with your health care team. If you have any questions, you can ask your study doctor for more explanation.

This study is being carried out under the sponsorship of Levine Cancer Institute (LCI). Novocure is the company that developed Optune<sup>TM</sup> that will be used in this study.

### WHY IS THIS STUDY BEING DONE?

The main purpose of this study is to see if adding Optune<sup>TM</sup> and bevacizumab to the standard medical treatment plan for GBM will increase the number of people who are alive after 12 months.

### HOW MANY PEOPLE WILL TAKE PART IN THE STUDY?

A total of approximately 46 subjects will take part in this study and will be enrolled in two groups. In the first group, 22 subjects will be enrolled. If adding Optune<sup>TM</sup> and bevacizumab to regular care shows an improvement in survival in the first group, the study will continue and will enroll the additional group of 24 patients. If adding Optune<sup>TM</sup> and bevacizumab to regular care does not show an improvement in survival in the first group, the 24 additional subjects will not be enrolled.

### **HOW THE STUDY WORKS**

### Before you begin the study (Pre-Study Treatment):

You will need to have the following tests and procedures done to determine if you can be in the study. These exams, tests, and procedures are part of regular cancer care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

- Demographics and medical history
- Physical and neurological (pertaining to the nervous system) examinations; including vital signs (heart rate, blood pressure, temperature) and height/weight measurements
- Performance status assessments (assesses daily living abilities)
- Magnetic Resonance Imaging (the use of magnetic waves to look at the soft tissues of the body) (MRI) of your brain
- Pregnancy test if able to get pregnant
- Documentation of any side effects you are experiencing
- Blood work for blood counts and biochemistry (electrolytes [salts or chemicals in the blood] and kidney and liver functions).

### During study treatment (Intervention):

If the exams, tests, and procedures show that you can be in the study, and you choose to take part, then you will receive the investigational treatment, Optune<sup>TM</sup> and bevacizumab, in addition to the standard medical treatment for newly diagnosed GBM

Ashley Sumrall, MD

patients. The current standard medical treatment typically begins with radiation therapy, along with the chemotherapy drug TMZ. You will first receive radiation therapy for five days each week for a total of six weeks. During this time, you will also take the oral study drug (pill) TMZ daily for six weeks and receive the intravenously injected (IV) drug BEV every two weeks, for approximately six weeks. At the end of this initial six week period, you will continue BEV every two weeks. After about four weeks, you will resume TMZ (daily on days 1-5 of each cycle) and continue BEV (every two weeks) for twelve cycles. A cycle is 28 days.

At this time, you will also begin study treatment with Optune<sup>TM</sup>. You will be asked to shave your head and wear the device for at least 18 hours a day (on average) for twelve months. While you are wearing the device, insulated transducer arrays (a ceramic disc coated with gel) will be attached to your shaved scalp using a bandage-like adhesive. The insulated transducer arrays produce alternating electric fields that interfere with the rapid cell division of cancer cells. At the end of the twelve months, you will stop wearing the device, but may continue to receive TMZ and BEV therapy at your physician's discretion.

During the study, you will need the following exams, tests, and procedures. Most of these exams, tests, and procedures are part of regular cancer care:

- Physical and neurological examinations
- Performance status assessment
- MRI scan of your brain
- Documentation of any side effects you experience
- Blood work for blood counts and biochemistry

### After you complete study treatment (End of Study Treatment visit):

When your study doctor discontinues your treatment with Optune<sup>TM</sup> (or if applicable, at the time of your doctor's decision that you will not be able to have the device placed) you will return for your End of Treatment visit. During this visit, the following procedures and tests will be done:

- Physical and neurological examinations; including vital signs (heart rate, blood pressure, temperature)
- Performance status assessment
- Documentation of any side effects you have experienced from study treatment
- Blood work for blood counts and biochemistry

# Follow-up:

When you have completed your End of Study Treatment visit, you will enter the follow-up period. You will remain in the follow-up period for the rest of your life, until you choose to quit the study, or until your study doctor removes you from the study.

Ashley Sumrall, MD

For subjects who have Optune<sup>TM</sup> placed during the study, the following procedures and tests will be done monthly during follow-up:

- Physical and neurological examinations; including vital signs (heart rate, blood pressure, temperature)
- Performance status assessment
- MRI scan of your brain (approximately every 8 weeks or as clinically indicated)
- Documentation of any side effects you are experiencing from study treatment

For subjects who have Optune<sup>TM</sup> placed during the study who show evidence of cancer worsening, the procedures listed above will no longer be required for follow-up. The following will be done approximately every 3 months during follow-up:

• Phone contact by the study team if you have not been seen by a healthcare provider around the time your 3-month follow-up contact is due

For subjects who are not able to have Optune<sup>TM</sup> placed during the study, you will be followed to monitor for side effects until 30 days after your last dose of study treatment. After this follow-up period has been completed, you will be removed from the study and will not be required to have any more follow-up visits for the purposes of the study.

### YOUR ROLE IN THE STUDY

Taking part in a research study can be an inconvenience to your daily life. Please consider the study time commitments and responsibilities as a research subject when you are deciding to take part. Your responsibilities as a study subject include the following:

- Tell the truth about your medical history and current conditions.
- Tell the study doctor if you have been in a research study in the last 30 days or are in another research study now.
- Tell the study doctor about any problems you have during the study.
- Use the study drug and study device as directed by the study doctor and study staff.
- Do not share the study drug and study device with anyone else. Keep the study drug and study device out of the reach of children and persons of limited capacity to read or understand.
- The study doctor or study staff will talk to you about any food or medicines that you should not take while in this study.
- Use care when driving or using machinery while you are taking the study drug and using the study device.
- Accurately fill out your TMZ pill diary and return it.

Ashley Sumrall, MD

### **RISKS**

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. However, doctors don't know all the side effects that may happen. Side effects may be mild or very serious. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after you stop taking the drugs, change the position of the transducer arrays or stop wearing the device. In some cases, side effects can be serious, long lasting, or may never go away. A severe side effect rarely may be life threatening. Although the risk of death is low, you should tell your study doctor immediately if you experience any side effects.

All side effects will be treated in the best way possible and this may involve anti-nausea medications, hospitalization to receive antibiotics (medications to fight infections), platelet (small cells in the blood that stop bleeding) transfusions (getting blood cells from another person), stool softeners or laxatives, and steroids or antihistamines for allergic reactions. There are guidelines for reducing the doses of chemotherapy drugs or eliminating them altogether should you experience serious or intolerable side effects. To avoid potential drug interactions, you should consult your physician or pharmacist before taking any new medications, including over the counter (non-prescription) medications.

This study has several risks. First, it is possible that you will get the new study treatment but do less well than you have been doing. Second, because the study treatment is new, we may not yet know all the side effects and something unexpected could happen. The following known side effects of radiation, Optune<sup>TM</sup>, BEV and TMZ are listed below.

### Risks and side effects of Radiation:

### Likely

- Scalp redness or soreness
- Hair loss, which may be temporary or permanent
- Ear/ear canal reactions, possibly resulting in a short-term hearing loss
- Fatigue (tiredness)
- Lethargy (sleepiness)
- Difficulty with concentration
- Temporary aggravation of brain tumor symptoms such as headaches, seizures, or weakness

# Less Likely

- Neurocognitive (thinking and understanding) problems, including memory deficits (loss), that could be permanent
- Permanent hearing loss
- Cataracts (clouding of the lens of the eye)
- Behavioral change

Ashley Sumrall, MD

- Nausea
- Vomiting
- Temporary worsening of existing neurological deficits, such as decreased vision, drowsiness, and weakness of your arms and legs
- Endocrine problems causing abnormalities in the level of some hormones (chemicals in the body) related to changes to the pituitary gland (produces hormones)
- Dry mouth or altered (changed) taste

### Rare but Serious

- Severe local damage to normal brain tissue, a condition called necrosis (tissue injury)
- Radiation necrosis can mimic recurrent (happens again) brain tumor and may require surgery for diagnosis and treatment
- Injury to the eyes with the possibility of blindness
- Development of other tumors (either benign [non-cancerous] or malignant [cancerous])

# Risks and side effects of Optune<sup>TM</sup>:

# Likely

- Local heat and tingling "electric" sensation beneath the transducer array
- Mild to moderate contact dermatitis (sore, red or inflamed skin) underneath the device

### Less Likely

- Skin irritation or skin breakdown
- Infection at the sites of transducer array contact with the skin
- Open sore, ulceration or blisters underneath the transducer arrays
- Headache
- Fatigue
- Weakness
- Convulsions
- Thinking changes

### Rare but Serious

• None previously reported

# Risks and side effects of Bevacizumab (BEV):

### Likely

- Loss of the normal functioning of the ovaries in a woman that can result in temporary or permanent menopause; the impact on fertility is unknown
- High blood pressure

### Less Likely

- Lack of enough red blood cells (anemia)
- Fever associated with dangerously low levels of a type of white blood cell (neutrophils)
- Fast heartbeat that usually starts in an area located above the ventricles
- Feeling of spinning or whirling
- Belly pain
- Inflammation (swelling and redness) of the large bowel (colon)
- Constipation
- Diarrhea
- Heartburn
- Bleeding in some organ(s) of the digestive tract
- Blockage in an organ(s)/part(s) of the digestive tract
- Partial or complete blockage of the small and/or large bowel
- Irritation or sores in the lining of the mouth
- Nausea or the urge to vomit
- Vomiting
- Fatigue or tiredness
- Reaction that can occur during or following infusion of the drug. The reaction may include fever, chills, rash, low blood pressure, and difficulty breathing
- Chest pain that is not heart-related
- Pain
- Allergic reaction by your body to the drug product that can occur immediately or may be delayed. The reaction may include hives, low blood pressure, wheezing, swelling of the throat, and difficulty breathing
- Infection
- Infection (collection of pus) around the rectum
- Premature opening of a wound along surgical stitches after surgery
- Increased blood level of a liver enzyme (ALT/SGPT)
- Increased level of a liver or bone enzyme (alkaline phosphatase)
- Increased blood level of a liver enzyme (AST/SGOT)
- Increased blood level of a liver pigment (bilirubin) often a sign of liver problems
- Increased blood level of a heart muscle protein (troponin I) indicating damage to the heart muscle
- Decreased number of a type of white blood cell (neutrophil/granulocyte)

Ashley Sumrall, MD

- Weight loss
- Decrease in the total number of white blood cells (leukocytes)
- Loss of appetite
- Joint pain
- Abnormal changes in the growth plate that may affect the growth of long bones in very young children. This side effect appeared to be reversible after the treatment was stopped but has not been assessed with long-term use of the bevacizumab drug.
- Muscle pain
- Destruction or death of jawbone
- Dizziness (or sensation of lightheadedness, unsteadiness, or giddiness)
- Headache or head pain
- Inflammation (swelling and redness) or degeneration of the peripheral nerves (those nerves outside of brain and spinal cord) causing numbness, tingling, burning
- Fainting
- Blood in the urine
- More protein leaking into the urine than usual, often a sign of kidney disease
- Bleeding in the vagina
- Stuffy or runny nose, sneezing
- Cough
- Shortness of breath
- Nose bleed
- Hoarseness
- Itching
- Skin rash with the presence of macules (flat discolored area) and papules (raised bump)
- Hives
- Formation of a blood clot that plugs the blood vessel; blood clots may break loose and travel to another place, such as the lung

### Rare but Serious

- Damage of or clots in small blood vessels in the kidney that can cause complications, some of which are serious including abnormal destruction of red blood cells (hemolysis) or platelets (that help to clot blood) and kidney failure
- Collection of signs and symptoms that indicate sudden heart disease in which the heart does not get enough oxygen. Sudden symptoms such as chest pain, shortness of breath, or fainting could indicate heart disease and should be reported right away.
- Heart failure: inability of the heart to adequately pump blood to supply oxygen to the body
- Decrease in heart's ability to pump blood during the "active" phase of the heartbeat (systole)
- Heart attack caused by a blockage or decreased blood supply to the heart
- Irregular heartbeat resulting from an abnormality in the one of the lower chambers of the heart (ventricle)

Ashley Sumrall, MD

- Ventricular fibrillation: irregular heartbeat that involves the lower chambers of the heart (ventricles) that results in uncoordinated contraction of the heart; life threatening and potentially fatal, needing immediate attention
- Gastrointestinal fistula: Abnormal hole between an organ of the digestive tract and another organ or tissue
- Gastrointestinal perforation: A tear or hole in the stomach or gut that can lead to serious complications and may require surgery to repair
- Sore (ulcer) somewhere in the digestive tract
- Serious, life-threatening allergic reaction requiring immediate medical treatment by your doctor. The reaction may include extremely low blood pressure, swelling of the throat, difficulty breathing, and loss of consciousness.
- Leakage from stomach due to breakdown of an anastomosis (surgical connection of two separate body structures)
- Bleeding in the brain
- Stroke caused by decreased blood flow to the brain
- Abnormal changes in the brain that can cause a collection of symptoms including headache, confusion, seizures, and vision loss associated with MRI imaging findings (RPLS)
- Sudden decrease of kidney function
- A condition in which the kidneys leak a large amount of protein into the urine that can cause complications including swelling and kidney failure
- Abnormal hole between part of the urinary system and another organ or tissue
- Abnormal hole between the vagina and another organ or tissue
- Abnormal hole between the lower breathing tube and the body cavity that surrounds the lungs
- Bleeding from the lungs
- Hole in the wall that separates the nostrils of the nose
- Abnormal hole between the breathing tube (windpipe) and the tube that goes from mouth to stomach through which food passes (esophagus). This is life-threatening and potentially fatal.
- Blockage or narrowing of a blood vessel (artery) that can cause damage or loss of function including a heart attack or stroke

# Risks and side effects of Temozolomide (TMZ):

### Likely

- Nausea and/or vomiting
- Decreased appetite
- Headache
- Constipation
- Drowsiness/Fatigue
- Inability to sleep

Ashley Sumrall, MD

### Less Likely

- Decrease in blood counts that may cause infection, bleeding, and bruising
- Diarrhea
- Fever
- Sores in your mouth
- Rash
- Elevated liver enzymes (chemicals in the liver) [reversible]
- Swelling in your arms and legs
- Memory loss
- Itchiness
- Increased need to urinate
- Weakness
- Back pain
- Dizziness
- Tingling/burning in your arms and legs
- Anxiety
- Depression
- Stomach pain

### Rare but Serious

- Decreased ability to carry out daily activities
- Convulsions
- Weakness on one side of your body
- Abnormal coordination
- Paralysis (inability to move)
- Myelodysplastic syndrome (problem with the bone marrow [soft tissue inside the bone] that causes decreased production of red cells, white cells, or platelets that can sometimes turn into blood cancer)

### Women Who Can Get Pregnant or Are Breastfeeding

You may not take part in this study if you are breastfeeding, are pregnant, think that you may be pregnant, or are trying to get pregnant. If you are pregnant or breastfeeding, there may be risks to you and the baby that are not known at this time. Women who can get pregnant will be tested for pregnancy during the study.

You must avoid getting pregnant in order to take part in this research study. You should not have sexual intercourse or you should use a method of birth control that is acceptable to you, the study doctor, and the sponsor during the study and six months after completion of the study treatment.

Ashley Sumrall, MD

It is important for you to tell the study doctor at once if you get pregnant or think that you might be pregnant while you are in the research study. If this happens, the study doctor will discuss with you what you should do. If you get pregnant, you will be asked to stop taking part in the study. You may also be asked questions about your pregnancy and the baby.

### Men

The effects of BEV and TMZ on male sperm is unknown. In rare cases, drugs may damage sperm in ways that affect a child that is fathered. Affected sperm may be present in the semen for about 2 months. In this study, however, it is recommended that males are to avoid fathering a child for 6 months after the last dose of the study treatment.

You should not have sexual intercourse or you should use a method of birth control that is acceptable to you, the study doctor, and the sponsor. If you think that you have gotten a woman pregnant, you must tell the study doctor at once. If your partner gets pregnant during the study, you may be asked questions about the pregnancy and the baby.

### Blood Draw/IV/Catheter Insertion Risks

You may have pain or bruising at the site where the blood is drawn or IV/catheter is inserted. You may feel faint. An infection at the site of the blood draw or IV/catheter insertion is possible.

### Allergic Reaction Risks

As with taking any drug, there is a risk of allergic reaction. If you have a very serious allergic reaction, you may be at risk of death. Some symptoms of allergic reactions are:

- Rash
- Wheezing and difficulty breathing
- Dizziness and fainting
- Swelling around the mouth, throat or eyes
- A fast pulse
- Sweating

Please seek treatment immediately and tell the study doctor and study staff if you have any of these symptoms, or any other side effects, during the study.

If you have problems that might be related to the drugs or device, you study doctor may remove you from the study.

Ashley Sumrall, MD

### **EXCLUSION CRITERIA**

The following conditions may prevent you from enrolling on this study. This is not a complete list. Your study doctor will review your medical record and the complete list of exclusion criteria in the study to see if they are applicable to you.

- Enrolled in another clinical treatment trial
- Pregnant or breast-feeding
- Any other cancer within the past 2 years aside from the following: localized basal cell or squamous cell carcinoma of the skin, cancer requiring hormonal therapy alone for management, and/or an early stage cancer that was cured by surgery
- Significant health conditions which would prevent you from taking temozolomide
- Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
- History of an allergy to bevacizumab, temozolomide, DTIC, or hydrogel
- Unwillingness to wear Optune<sup>TM</sup> for an average of 18 hours per 24 hours
- New York Heart Association (NYHA) Grade II or greater congestive heart failure
- History of heart attack or unstable angina (chest pain) within the last 6 months
- History of stroke or transient ischemic attack (TIA) within the last 6 months
- Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within the last 6 months
- History of coughing up blood within the last month
- Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to 1<sup>st</sup> bevacizumab infusion or anticipation of need for major surgical procedure during the course of the study
- Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
- History of abdominal fistula, gastrointestinal perforation within the last 6 months
- Serious, non-healing wound, active ulcer, or untreated bone fracture

### WILL I BENEFIT FROM PARTICIPATING IN THIS STUDY?

This study may or may not improve your condition. The information gained from your participation may benefit others with your condition.

### WHAT OTHER CHOICES DO I HAVE IF I DO NOT TAKE PART IN THIS STUDY?

Your other choices may include:

- Getting treatment or care for your brain tumor without being in a study; this could include bevacizumab plus the standard medical therapy (radiation plus temozolomide).
- Taking part in another research study

Ashley Sumrall, MD

• Getting no treatment other than close observation and follow-up

### WHAT ARE THE COSTS OF TAKING PART IN THIS STUDY?

Novocure, the manufacturer of Optune<sup>TM</sup>, will attempt to seek reimbursement from your insurance company for use in this clinical trial. Depending on your insurance company, you may have coverage for Optune<sup>TM</sup> while participating in this clinical trial. If your insurance company does not provide coverage for Optune<sup>TM</sup> or your out of pocket financial cost share would be unaffordable, you may be eligible for financial assistance. It is recommended that you contact Novocure prior to signing this consent at

You and/or your health plan/insurance will need to pay for some or all of the costs related to your radiation therapy and chemotherapy treatment (bevacizumab and temozolomide).

Certain tests and examinations will need to be done regularly to monitor your safety and to measure the effects of chemotherapy and Optune<sup>TM</sup>. These tests include physical exams, scans, urine tests, and blood tests. Costs for these tests and examinations will be billed to you and/or your health plan/insurance. The use of medications or other types of treatment to help control side effects you might have could also result in added costs to you and/or your health plan/insurance.

You will not receive payment for taking part in this study. For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this web site. Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

### STUDY STAFF PAYMENT/FINANCIAL DISCLOSURE

The manufacturer of Optune<sup>TM</sup>, Novocure, will give and has given the study doctor, Dr. Ashley Sumrall, money or other benefits to be used for the cost of conducting the study.

### WHAT HAPPENS IF I AM INJURED BECAUSE I TOOK PART IN THIS STUDY?

If you become ill or are hurt while you are in the study, get the medical care that you need right away.

In the event that you are harmed as a result of your participation in this study, inform your study doctor immediately so you can access medical treatment. You and/or your health plan will be charged for this treatment in the usual manner. The study will not pay for standard medical treatment.

You still have the right to make a claim through the legal system even if you sign this form, accept medical care, or accept payment for medical expenses.

Ashley Sumrall, MD

We will tell you about new medical findings that may affect your willingness to continue in the study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a> as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

### **CONFIDENTIALITY**

The records of this study will be kept private. In any sort of report we might publish, we will not include any information that will make it possible to identify a patient. Your record for this study may, however, be reviewed and/or photocopied by the drug/device manufacturer/sponsor, by Carolinas HealthCare System, or by representatives of the Food and Drug Administration or other government agencies. To that extent, confidentiality is not absolute.

To ensure that your information collected for this study will be kept private, your name will not be used whenever possible. A code will be used instead of your name. All of your study data will be kept in a secure location.

### AUTHORIZATION TO DISCLOSE HEALTH INFORMATION

If you wish to take part in this clinical study, you will be asked to sign this consent form. It allows the study sponsor and the study investigator to collect, process and pass on to the sponsor organizations any relevant personal health information collected from you during the study. These are activities routinely carried out during all clinical studies.

You have been told that personal information about you (including sensitive personal health information, such as your medical history and your racial/ethnic origin if relevant to the study) will be reviewed, collected on a computer database, stored in electronic or manual files, audited, and/or otherwise processed by:

- the study doctor and study staff,
- the study sponsor and/or its associated companies, Levine Cancer Institute, Novocure
- regulatory or other governmental authorities of the United States and other countries,
- other persons authorized by the study sponsor,
- Carolinas HealthCare System employees,
- other persons or agencies as required by law or allowed by federal regulations.

You have been told that your personal data are being collected and processed to:

- check your suitability to take part in the study,
- monitor your treatment with the study drugs/device,

Ashley Sumrall, MD

- compare and pool study treatment results with those of other subjects in clinical studies,
- support the development of the study drugs,
- support the licensing application for regulatory approval of the study drugs or device in the world
- support the marketing, distribution, sale and use of the study drugs or device anywhere in the world.

You have been told that your personal information may be processed within the U.S. or elsewhere in the world or transferred to or from the U.S. for review, processing and/or storage by an associated company or a carefully selected third-party organization. By signing this document, you explicitly consent to the transfer of your personal information, including sensitive personal information, collected during this clinical study, for review, processing and/or storage. Your personal health information may be further shared by the groups above. If shared by them, the information will no longer be covered by the Privacy Rule. However, the groups are committed to keeping your personal health confidential.

You may refuse this authorization to transfer your personal information. If you choose not to agree to this authorization, you might be ineligible to participate in the study. If you decide not to sign this authorization, that will not harm your relations with your doctors or with Carolinas HealthCare System.

You have the right to inspect your medical record at any time. Your research record may be unavailable until the conclusion of the study. At that point, it will be available. Please speak with the study doctor if you desire to access your record.

You have been told whenever your personal information is processed; it will be kept confidential and secure, to the best of our ability. It will be used only for the purpose for which it was collected.

This Authorization does not have an expiration date. You have been told that according to the guidelines for good clinical practice, the study investigator and sponsor will keep your personal information for at least 6 years. If you do not withdraw this Authorization in writing, it will remain in effect indefinitely. If you wish to revoke authorization to use your personal information, you will notify the study doctor in writing at the address and telephone number listed on the first page of this form. Some of the data obtained from your record prior to your revocation may still be used if considered necessary for the study.

# GETTING ANSWERS TO YOUR QUESTIONS ABOUT THE STUDY

You can ask questions about this consent form or the study (before you decide to start the study or at any time during the study). Questions may include:

- Who to contact in the case of a research-related injury or illness
- Any payment for being in the study
- Your rights and your responsibilities as a study subject
- Other questions

Contact the study doctor or study staff at Carolinas HealthCare System with any questions or concerns. Their telephone number is printed on the first page of this form. If you have any questions or complaints about your rights as a research subject, contact:



Please reference the following number when contacting the Study Subject Adviser: <u>Pro00010270</u>.

If you seek emergency care, or if hospitalization is required, please inform the treating doctor that you are participating in a clinical trial.

If any new information becomes available during the course of this study that may affect your willingness to participate, you will be informed.

### BEING A STUDY VOLUNTEER AND WITHDRAWING FROM THE STUDY

Your participation in this study is completely voluntary. You should feel under no pressure to be in the study. If you decide not to be in the study that will not in any way harm your relations with your doctors or with Carolinas HealthCare System. You are free to stop being in the study if you change your mind after entering it. This would not harm your relations with your doctors or Carolinas HealthCare System.

- You may always say no. You do not have to take part in the study.
- If you start a study, you may stop at any time. You do not need to give a reason.
- If you do not want to be in a study or you stop the study at a later time, you will not be penalized or lose any benefits.

Ashley Sumrall, MD

• If you stop, you should tell the study staff and follow the instructions they may give you.

Your part in the research may stop at any time for any reason, such as:

- The sponsor or the study doctor decides to stop the study.
- The sponsor or the study doctor decides to stop your part in the study for your safety.
- You need additional medicine.
- You do not follow the study rules.
- You have a new injury or illness.
- You decide to stop.

You may be asked to stop the study even if you do not want to stop.

# STATEMENT OF CONSENT

| Thave read this form and its contents were explained to a<br>the purposes listed above. All of my questions were answ<br>signed and dated copy of this form for my records. I am<br>signing this form. | wered to my satisfaction. 1 | will receive a |
|---|---|---|
| | // | |
| Signature of Research Subject | Date | Time |
| Printed Name of Research Subject | | |
| STATEMENT OF PERSON EXPLAINING CONSTITUTE IN THE STATEMENT OF PERSON EXPLAINING CONSTI | ourpose of the above study<br>s research study. I have be | |
| , | / / | |
| Signature of Person Explaining Consent | //<br>Date | Time |
| Printed Name of Person Explaining Consent | | |